CLINICAL TRIAL: NCT03362515
Title: Treatment of Post-Operative Sinonasal Polyposis With Topical Furosemide
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated prematurely due to low enrollment numbers and the development of better drugs to treat polyps (ie. Biologics) which were not available when the study began.
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17D.264
Record Dates: First submitted 2017-11-28; First posted 2017-12-05 (Actual); Results first posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Nasal Polyps
MeSH Terms: conditions — Nasal Polyps | interventions — Furosemide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Furosemide (Experimental)
  Interventions: Drug: Furosemide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Furosemide — furosemide
  Arms: Furosemide
Drug: Placebo — placebo
  Arms: Placebo

SUMMARY:
Prior studies have suggested that topical furosemide may reduce the recurrence of sinonasal polyposis following sinus surgery. This project aims to further investigate that claim through a blinded randomized controlled clinical trial following patients who undergo functional sinus surgery for chronic rhinosinusitis with sinonasal polyposis by randomly assigning participants to receive topical furosemide versus placebo nasal spray for 2 months post operatively. Outcomes would be compared at 6 months through endoscopic grading scores using Lund Kennedy and Meltzer scores as well as Sino-Nasal Outcome Test (SNOT-22) scores to measure the rate and degree of recurrence and impact on symptoms in the treatment group versus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic rhinosinusitis and sinonasal polyposis who are candidates for functional endoscopic sinus surgery

Exclusion Criteria:

* Hypersensitivity to furosemide or sulfonamides
* pregnancy
* history of tinnitus
* history of sensorineural hearing loss
* poorly controlled diabetes
* current diuretic therapy
* known electrolyte disorder
* currently taking aminoglycosides
* BUN and creatinine levels out of the normal range
* history of renal disease
* allergy to sulfonamides

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Department of Otolaryngology, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Furosemide | Placebo
Started | 9 | 9
Completed | 6 | 6
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Furosemide | Placebo | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Polyp Recurrence
Description: Nasal and paranasal polyposis based on endoscopic grading through Lund Kennedy score to measure the rate and degree of recurrence.
Time Frame: 6 months
Population: This data was not collected and therefore no data analysis was done due to the study being terminated early secondary to 1) low enrollment due to the emergence of better medical alternatives to treat polyps (ie. Biologics) which made using furosemide not useful and 2) COVID.
Arm/Group | Furosemide | Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Polyp Recurrence
Description: Nasal and paranasal polyposis based on endoscopic grading through Meltzer score to measure the rate and degree of recurrence.
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | Furosemide | Placebo
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Polyp Recurrence
Description: Nasal and paranasal polyposis based Sino-Nasal Outcome Test (SNOT-22) scores to measure impact on symptoms.
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | Furosemide | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Furosemide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 1/9 | 3/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Furosemide (N=9) | Placebo (N=9)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
increased headaches (General disorders) | 0 (0) | 1 (1)
burning sensation in throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-10): https://cdn.clinicaltrials.gov/large-docs/15/NCT03362515/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/15/NCT03362515/ICF_001.pdf